CLINICAL TRIAL: NCT06076629
Title: Acute Health Effects of Low Temperature Exposure in Healthy Young Adults: A Randomized Controlled Study
Brief Title: Acute Health Effects of Low Temperature Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FDUEH-9
Record Dates: First submitted 2023-09-08; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular System; Respiratory System; Cognitive Function
Keywords: Low temperature; Randomized controlled trial; Cardiopulmonary effects; Cognitive function
MeSH Terms: interventions — Cold Temperature; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low temperature (16#) group (Experimental): Subjects in exposure group will be exposed to low temperature (16#) for about 2 hours in a chamber.
  Interventions: Other: Low temperature (16#) group
- Moderate temperature (22#) group (Sham Comparator): Subjects in exposure group will be exposed to moderate temperature (22#) for about 2 hours in a chamber.
  Interventions: Other: Moderate temperature (22#) group

INTERVENTIONS:
Other: Low temperature (16#) group — The exposure group will be exposed to low temperature (16#) in a chamber for about 2 hours, resting during the whole periods.
  Arms: Low temperature (16#) group
Other: Moderate temperature (22#) group — The exposure group will be exposed to thermoneutral temperature (22#) in a chamber for about 2 hours, resting during the whole periods.
  Arms: Moderate temperature (22#) group

SUMMARY:
This is a randomized controlled human exposure crossover study. Investigators aims to assess the acute effects of low temperature exposure and the underlying mechanisms.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled human exposure crossover study among about 50 healthy young adults in Shanghai, China. Each subject will be exposed twice: once to the low temperature (16#) and once to the moderate temperature (22#) in a chamber for about 2-2.5 hours. During the exposure session, each subject will be requested to rest. Health examinations will be conducted immediately prior to exposure (within 1 hour before the exposure session), during the period of exposure, and after exposure (within 2 hours after the exposure session). Health examinations include spirometry, Holter monitoring, blood pressure tests, cognitive function tests, symptom questionnaires, and magnetic resonance imaging. Investigators plan to collect blood, urine, exhaled breath condensate, and oropharyngeal swabs samples.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during the study period;
* Body mass index > 18.5 and ≤ 28;
* Right-handed;
* Receiving or having received higher education;
* With the ability to read and understand Chinese smoothly.

Exclusion Criteria:

* Smoking and alcohol abuse;
* Current drug and dietary supplements intake;
* Subjects with allergic diseases, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular diseases, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory diseases, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic diseases, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects who have a history of major surgery due to cardiovascular, cerebrovascular, respiratory, or neurological diseases;
* Subjects with neurologic disorders, such as stroke, traumatic brain injury, epilepsy, and schizophrenia;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Subjects with color vision disabilities.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability Parameters | Volunteers will be asked to wear electrographic Holter monitors for 24 hours from 1:00 P.M. at the day of intervention to 1:00 P.M. at the next day.
  Investigators plan to measure heart rate variability (HRV) parameters (e.g., SDNN, PNN50, LF, HF)
Blood Pressure | Blood pressure will be examined before exposure and immediately after the exposure session
  The changes of systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be measured.
Forced vital capacity | Lung function will be examined before exposure and half an hour after the exposure session
  Investigators plan to measure forced vital capacity (FVC) by spirometry
Forced expiratory volume in one second | Lung function will be examined before exposure and half an hour after the exposure session
  Investigators plan to measure forced expiratory volume in one second (FEV1) by spirometry.
Maximal mid-expiratory flow | Lung function will be examined before exposure and half an hour after the exposure session
  Investigators plan to measure maximal mid-expiratory flow (MMEF) by spirometry.
Results of Stroop Tests | The tests will be conducted before exposure and immediately after the exposure session
  Investigators plan to measure the changes of cognitive function using Stroop Test.

SECONDARY OUTCOMES:
Changes of skin temperature | Skin temperature will be examined from 1:00 P.M. to 4:30 P.M. at the day of intervention
  The changes of wrist skin temperature will be measured
Results of simple reaction time | Simple reaction time will be examined before exposure and immediately after the exposure session
  Investigators plan to measure the changes of cognitive function using visual simple reaction time test.
Results of visual memory | Visual memory will be examined before exposure and immediately after the exposure session
  Investigators plan to measure the changes of cognitive function using visual memory test. Every level, a number of tiles will flash white. The participants will be required to memorize them, and pick them again after the tiles are reset. Higher levels refer to better visual memory.
Activated brain regions demonstrating brain activity related to the low temperature exposure | MRI will be examined 1 hour after the exposure session
  Investigators plan to conduct magnetic resonance imaging (MRI) after exposure. The MRI data will be processed through Data Processing and Analysis for Brain Imaging (DPABI) sofrware to obtain brain activity parameters, such as fractional amplitude of low-frequency fluctuation (fALFF). Brain regions that change after exposure between the two groups would be further idenfitied.
Changes in cerebral hemodynamics demonstrating brain activity related to the low temperature exposure | fNIRS will be examined before exposure and immediately after the exposure session
  Investigators plan to conduct functional near-infrared spectroscopy (fNIRS) to measure the changes in oxygenated hemoglobin and deoxygenated hemoglobin after exposure. Matlab would be applied to process data and evaluate the changes in cerebral hemodynamics associated with low temperature exposure

OTHER OUTCOMES:
Differences in metabolites detected in blood between the two exposures | Blood will be collected 1 hour after the exposure session
  The differentially expressed metabolites in blood related to low temperature exposure will be detected by maspectrometry-based non-targeted metabolomics.
Differences in protein levels detected in blood between the two exposures | Blood will be collected 1 hour after the exposure session
  The differentially expressed proteins in blood related to low temperature exposure will be detected by non-targeted proteomics.
Differences in DNA methylation levels detected in whole-blood between the two exposures | Blood will be collected 1 hour after the exposure session
  Genome-wide DNA methylation in whole-blood were detected. The study is to identify differential CpG loci after low temperature exposure
Changes of the scores of thermal sensation questionnaires | The questionnaires will be conducted before exposure and immediately after the exposure session
  Changes of scores of thermal sensation questionnaires which ranged from -5 to 5. Zero score refers to the thermal comfort sensation. Higher scores refer to more uncomfortable sensations of hot. Lower scores refer to more uncomfortable sensations of cold.
Changes of scores of symptoms questionnaires | The questionnaires will be conducted before exposure and immediately after the exposure session
  Changes of scores of respiratory and cardiovascular symptoms questionnaires which ranged from 0 to 5. Zero score refers to no symptoms, and higher scores refer to more severe symptoms.
Change in C reactive protein (CRP) concentrations | Blood will be collected 1 hour after the exposure session
  Change in the concentrations of C reactive protein in blood.
Changes of facial secreted sebum composition | Facial sample will be collected half an hour after the exposure session
  Investigators plan to collect facial secreted sebum composition using Sebutape. The differential facial secreted sebum composition between the two groups would be further evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, PhD, Study Director — Department of Environmental Health, School of Public Health, Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No